CLINICAL TRIAL: NCT06976268
Title: A Phase 2/3, Double-Blind, Placebo-Controlled Study of BHV-8000 in Participants With Early Parkinson's Disease
Brief Title: A Study to Determine if BHV-8000 is Effective, Safe and Tolerable as a Treatment for Adults Living With Early Parkinson's Disease
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Biohaven Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Organization: Biohaven Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BHV8000-301; 2025-521113-13-00 (EU CTIS Number)
Record Dates: First submitted 2025-05-09; First posted 2025-05-16 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease
Keywords: Early Parkinson's Disease; Parkinson's Disease; Early onset Parkinson's Disease; treatment naiive early Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BHV-8000 10 mg (Experimental)
  Interventions: Drug: BHV-8000
- BHV-8000 20 mg (Experimental)
  Interventions: Drug: BHV-8000
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BHV-8000 — BHV-8000 10 mg. Participants will take blinded investigational product (IP) once daily
  Arms: BHV-8000 10 mg
Drug: BHV-8000 — BHV-8000 20 mg. Participants will take blinded investigational product (IP) once daily
  Arms: BHV-8000 20 mg
Drug: Placebo — Matching placebo taken once daily
  Arms: Placebo

SUMMARY:
A study to determine if BHV-8000 is efficacious, safe and tolerable in adults diagnosed with early Parkinson's disease.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female participants 40 to 85 years of age, inclusive, at the time of informed consent.
* Meet the diagnostic criteria for "Probable PD" as assessed on the Movement Disorder Society (MDS) Clinical Diagnostic Criteria for PD as assessed by the Investigator.
* Have a clinician-documented diagnosis of idiopathic PD with an onset within 2 years of the Screening Visit

Key Exclusion Criteria:

* Medical history indicating a Parkinsonian syndrome other than idiopathic PD, including, but not limited to, progressive supranuclear gaze palsy, multiple system atrophy, drug-induced Parkinsonism, essential tremor, or primary dystonia.
* Diagnosis of clinically significant central nervous system (CNS) disease other than PD.
* Participants who are current smokers (defined as smoking [in any form, e.g., tobacco smoke, electronic cigarettes, etc.] )
* Treatment with PD medication(s)
* Any other condition(s) that may compromise participant safety, interfere with study conduct, or jeopardize the potential proper interpretation of study results, in the opinion of the investigator.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Time to first qualifying worsening event on Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part II | Up to 48 Weeks
  To evaluate the efficacy of BHV-8000 compared to placebo. This objective is measured by assessing the time to prespecified worsening on MDS-UPDRS Part II (motor experiences of daily living per self-administered questionnaire). MDS-UPDRS Part II is a 52-point scale with a higher total score representing more severe disability.

SECONDARY OUTCOMES:
Change in Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III from Baseline to Week 48 | Baseline to Week 48
  To evaluate the efficacy of BHV-8000 compared to placebo. This objective is measured by assessing the change in MDS-UPDRS Part III (motor examination conducted by rater). MDS-UPDRS Part III is a 132-point scale with a higher total score representing a greater degree of motor impairment.
Change in Clinical Global Impression of Severity (CGI-S) from Baseline to Week 48 | Baseline to Week 48
  To evaluate the efficacy of BHV-8000 compared to placebo. This objective is measured by assessing the change in severity of a participant's illness as determined by the managing clinician. The CGI-S is a 7-point scale (1 - 7) with 7 representing the most extremely ill participants.
Change in DaT-SPECT scan from Baseline to Week 48 | Baseline to Week 48
  To evaluate the efficacy of BHV-8000 compared to placebo. This objective is measured by change in DaT-SPECT Striatal Binding Ratio (SBR) in the putamen (assessing the activity of the dopamine transporters). Reduced uptake of the radiotracer is indicative of a decreased number of dopamine-secreting cells and suggestive of disease progression.
Change in Parkinson's Disease Composite Score - Function (PARCOMS-Function) from Baseline to Week 48 | Baseline to Week 48
  To compare the efficacy of BHV-8000 compared to placebo. This objective is measured by changes in the Parkinson's Disease Composite Score - Function (PARCOMS-Function) score. The PARCOMS-Function is a composite of select items taken from the MDS-UPDRS Part II and the PDQ-39© (assessing ability to complete daily activities). The PARCOMS-Function is a 100-point scale (0 - 100) with higher scores representing greater dysfunction.
Number of Participants with Deaths, Serious AEs (SAEs), AEs Leading to Study Drug Discontinuation, and moderate or severe AEs | Baseline to Week 48
  To assess the safety and tolerability of BHV-8000. This objective will be measured by assessing the number of unique participants with deaths, SAEs, AEs leading to discontinuation, and moderate and severe AEs.
Number of participants with clinically significant laboratory abnormalities | Baseline to Week 48
  To assess the safety and tolerability of BHV-8000. This objective will be measured by assessing the number of unique participants with treatment-emergent Grade 3 and 4 laboratory abnormalities.

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Site-049, Birmingham, Alabama
  - Site-041, Los Angeles, California
  - Site-031, Farmington, Connecticut
  - Site-028, New Haven, Connecticut
  - Site-038, Atlantis, Florida
  - Site-017, Boca Raton, Florida
  - Site-051, Maitland, Florida
  - Site-027, Chicago, Illinois
  - Site-071, Boston, Massachusetts
  - Site-015, Farmington Hills, Michigan
  - Site-044, Chesterfield, Missouri
  - Site-005, New York, New York
  - Site-091, Portland, Oregon
  - Site-043, Round Rock, Texas
  - Site-007, Bellevue, Washington